CLINICAL TRIAL: NCT06210386
Title: Physiological Effects of Helmet vs. Facemask Noninvasive Ventilation in Acute Hypoxemic Respiratory Failure
Brief Title: Physiology of Helmet vs. Facemask Noninvasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5173-1
Record Dates: First submitted 2024-01-02; First posted 2024-01-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Crossover randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Helmet noninvasive ventilation (Experimental): 1-hour treatment with helmet noninvasive ventilation (PEEP 12 cmH2O + pressure support 10 cmH2O).
  Interventions: Device: Noninvasive ventilation
- Facemask noninvasive ventilation (facemask settings) (Active Comparator): 1-hour treatment with facemask noninvasive ventilation (PEEP 5 cmH2O + pressure support 10 cmH2O).
  Interventions: Device: Noninvasive ventilation
- Facemask noninvasive ventilation (helmet settings) (Active Comparator): 1-hour treatment with facemask noninvasive ventilation (PEEP 12 cmH2O + pressure support 10 cmH2O).
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: Noninvasive ventilation — noninvasive ventilation

SUMMARY:
The optimal noninvasive management of acute hypoxemic respiratory failure is debated. Helmet noninvasive ventilation may be more effective than facemask noninvasive ventilation for these patients. Putatitve benefits of helmet use are the possibility to apply significantly higher positive end-expiratory pressure without air leaks and with good patient's comfort.

In this randomized crossover study, the investigators will assess the physiological effects of helmet compared to facemask noninvasive ventilation, with the latter applied with different ventilator settings (similar to or different from helmet settings).

ELIGIBILITY:
Inclusion Criteria:

* Acute hypoxemic respiratory failure and PaO2/FiO2<200 mmHg
* PaCO2<45 mmHg
* Respiratory failure not caused by exacerbation of chronic pulmonary disease, cardiac failure or fluid overload

Exclusion Criteria:

* Pregnancy
* Contraindication to helmet or facemask noninvasive ventilation
* Contraindication to esophageal manometry
* Contraindication to electrical-impedance tomography monitoring
* Recent surgery involving the abdomen or the thorax
* Pneumothorax or documented barotrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Inspiratory effort | 1 hour
  negative deflection in esophageal pressure
End-expiratory lung impedance | 1 hour
  Electrical-impedance derived end-expiratory lung volume

SECONDARY OUTCOMES:
Tidal volume | 1 hour
  Electrical-impedance derived tidal volume size
Work of breathing | 1 hour
  Esophageal pressure simplified pressure-time product
Respiratory rate | 1 hour
  Respiratory rate per minute
Dynamic transpulmonary driving pressure | 1 hour
  Tidal change in transpulmonary pressure
Compliance | 1 hour
  Ratio of tidal volume to transpulmonary driving pressure
Dyspnea | 1 hour
  Dyspnea rated through a visual analog scale (ranging from 0 to 10, with representing most severe dyspnea) adapted for critically ill patients
Discomfort | 1 hour
  Device-related discomfort (ranging from 0 to 10, with representing most severe dyspnea) rated through a visual analog scale adapted for critically ill patients
Oxygenation | 1 hour
  PaO2/FiO2 ratio
Pendelluft extent | 1 hour
  Pendelluft extent, expressed in % of the total tidal volume
Corrected minute ventilation | 1 hour
  The product of tidal volume and respiratory rate, normalized to PaCO2. This value is expressed in Arbitrary units per minute divided by mmHg and is a proxy of dead space
Arteria Carbon dioxide tension | 1 hour
  PaCO2
Tidal volume distribution | 1 hour
  Tidal volume distribution, assessed with electrical impedance tomography in 4 regions of interest (ventral, mid-ventral, mid-dorsal, dorsal)

CONTACTS AND LOCATIONS:
Overall Officials: Domenico L. Grieco, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request